CLINICAL TRIAL: NCT01612078
Title: A Double-blind, Randomized and Placebo-controlled Study to Evaluate the Efficacy and Safety of L-threo-3,4-dihydroxyphenylserine (Droxidopa) on Orthostatic Hypotension Treatment in Hemodialysis Patients
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of Droxidopa on Orthostatic Hypotension Treatment in Hemodialysis Patients
Acronym: OH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSHDX1101
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Droxidopa, antihypotensive drug, tablet (Experimental)
  Interventions: Drug: Droxidopa
- placebo, tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Droxidopa — 200mg/tab 2tablets, po, three times a week
  Arms: Droxidopa, antihypotensive drug, tablet
Drug: Placebo — 200mg/tab, po, three times a week.
  Arms: placebo, tablet

SUMMARY:
Orthostatic hypotension is a major complication of hemodialysis and interferes with everyday activities in hemodialysis patients. Since information regarding the use of droxidopa in clinical trials relating to orthostatic hypotension of chronic hemodialysis patients is limited in Taiwan, this study is designed for evaluation the efficacy and safety profile of droxidopa on orthostatic hypotension treatment / prevention in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged great than 20 years of age
2. Patient with at least 3 month documented requirement of regular hemodialysis session
3. Patient with a decrease of 20 mmHg in SBP or 10 mmHg in DBP within 5 minutes of standing after the end of hemodialysis in at least 2 of 3 sessions during the screening period.
4. Subject with subjective complain of light headedness related to the orthostatic hypotension AND with a VAS score 4 in at least 2 of 3 sessions during the screening period.
5. Willing and able to comply with the study procedure and sign a written informed consent

Exclusion Criteria:

1. Female who is pregnant, lactating or planning to be pregnant within 3 months, or female of childbearing potential who is not using medically recognized method of contraception
2. Subject with closed angle glaucoma
3. Subject with severe hypertension
4. Subject with liver disorder
5. Subject with Hct great than 36%
6. Subject with confusion, hallucination, or delusion
7. Subject with severe disease which may limit survival during the study period, or confound the results of the study as judged by the investigator, such as hyperthyroidism, artery stenosis, severe lung disorders, severe asthma, chronic open angle glaucoma, uncontrolled diabetic gangrene
8. Subject who takes any anti-hypotensive drugs within 7 days prior to randomization, such as midodrine, etilefrine or amezinium
9. Subject who takes ephedrine, pseudoephedrine within 7 days prior to randomization
10. Subject who use of any investigational product within 4 weeks prior to randomization
11. Subject who requires blood transfusions within 3 months before screening, and are not suitable to participate the trial as judged by the investigator
12. Histories of hypersensitive to droxidopa
13. Histories of peripheral vascular disease, coronary artery disease and are not suitable to participate the trial as judged by the investigator
14. Histories of hemorrhage complication within 3 months before the screening visit, such as GI bleeding, intracranial bleeding or traumatic hemorrhage, and are not suitable to participate the trial as judged by the investigator
15. In investigator's opinion, subjects who are unlikely to adequately cooperate and follow the procedures

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in mean ΔSBP after hemodialysis | from Week 0 (visit 1-3) to Week 4 (visit 13-15)
  ΔSBP = supine SBP (right before standing up) - nadir standing SBP

SECONDARY OUTCOMES:
Adverse event,Serious adverse event | from week 0 to week 5

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Szu Wu, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan